CLINICAL TRIAL: NCT04745624
Title: Real World Use and Outcomes of VASCADE Closure Device Versus Manual Compression in Patients With Common Femoral Artery Disease: A Retrospective Comparison Study
Brief Title: Real World Use and Outcomes of VASCADE Closure Device Versus Manual Compression in Patients With CFA Disease
Acronym: VASCADE
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000028947
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Common Femoral Artery Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- manual compression cohort: Manual compression cohort: Patients who underwent coronary or peripheral angiograms via CFA access with moderate to severe stenosis were hemostasis was achieved via manual compression
- VASCADE cohort: VASCADE cohort: Patients who underwent coronary or peripheral angiograms via CFA access with moderate to severe stenosis were hemostasis was achieved via VASCADE device closure

SUMMARY:
To study the patient characteristics and outcomes associated with the real-world use of manual compression vs. vascular closure devices (VCDs) after common femoral artery (CFA) percutaneous access for coronary and endovascular interventions. An institutional procedural database, based on electronic medical record information will be abstracted to collect this information.

DETAILED DESCRIPTION:
The overall objective of the study will be to examine the safety and efficacy of the VASCADE closure device compared to manual compression (standard of care) to achieve hemostasis after endovascular procedures requiring access within a severely diseased CFA.

This study will be a retrospective single center review of 200 patients undergoing endovascular procedures utilizing vascular access within a severely diseased CFA between 2018 and 2020 at Yale New Haven Hospital. A random selection of patients undergoing hemostasis with manual compression (n = 100) and VASCADE vascular closure system (n = 100) will be conducted. The two groups will then be statistically compared with respect to 48-hour and 30-day safety and efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 5, 6 or 7 Fr access within the CFA
2. ACT < 300 seconds
3. Age 18 - 90 years old
4. Severe common femoral arterial disease Percent stenosis > 50, which will be core-lab adjudicated

Exclusion Criteria:

1. Ipsilateral CFA access within 30 days preceding or subsequent to the index case
2. Prior ipsilateral closure device use, other than VASCADE
3. High bleeding risk ACT > 300 or > 250 with IIb/IIIa inhibitor Plt < 50K INR > 1.7 on the day of procedure Inherent coagulopathy NOAC, warfarin, or lovenox administered within 24 hours of the procedure
4. Suspected intraluminal thrombus, dissection, pseudoaneurysm, hematoma, or AV Fistula

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective review of medical records and angiograms of patients who underwent coronary and peripheral angiograms at one institution. Patients with CFA stenosis will be identified by review of their access site angiograms. The method use for hemostasis, characteristics and outcomes will be abstracted via review of medical records.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Adequate hemostasis - (efficacy) | within an hour immediately after procedure
  No evidence of bleeding after device use
No complications after procedure - (safety) | early (48 hours)
  Early complications rates: bleeding, thrombosis, pseudoaneurysm, arterio-venous fistula, access site infection, mortality
No complications after procedure - (safety) | late (30-day)
  Late complications rates: bleeding, thrombosis, pseudoaneurysm, arterio-venous fistula, access site infection, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena-Hurtado, MD, Principal Investigator — Yale University; Kim Smolderen, Study Director — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bangalore S, Bhatt DL. Femoral arterial access and closure. Circulation. 2011 Aug 2;124(5):e147-56. doi: 10.1161/CIRCULATIONAHA.111.032235. No abstract available. PMID 21810667
- [Background] Noori VJ, Eldrup-Jorgensen J. A systematic review of vascular closure devices for femoral artery puncture sites. J Vasc Surg. 2018 Sep;68(3):887-899. doi: 10.1016/j.jvs.2018.05.019. Epub 2018 Jun 29. PMID 30146036
- [Background] Arora N, Matheny ME, Sepke C, Resnic FS. A propensity analysis of the risk of vascular complications after cardiac catheterization procedures with the use of vascular closure devices. Am Heart J. 2007 Apr;153(4):606-11. doi: 10.1016/j.ahj.2006.12.014. PMID 17383300